ClinicalTrials.gov ID: NCT03483961

Document: PXVX-CV-317-001 Protocol

Protocol Title: A Phase 2 Parallel-Group, Randomized, Double-Blind Study to Assess the Safety and Immunogenicity of PXVX0317 (Chikungunya Virus Virus-Like Particle Vaccine [CHIKV-VLP], unadjuvanted

or alum-adjuvanted)

Protocol Number: PXVX-CV-317-001

Protocol Version 4.0

Protocol Version Date: 22-May-2020 (Approval date: 27-May-2020)